CLINICAL TRIAL: NCT06809361
Title: Obesity Prevention Program for Overweight and Obese Adolescents
Brief Title: The Effectiveness of the Obesity Prevention Program Developed for Overweight and Obese Adolescents and Supported by Social Media Reminders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Adem SÜMEN, associate professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Obesity Prevention Program
Record Dates: First submitted 2025-01-27; First posted 2025-02-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Obesity Prevention
Keywords: Overweight adolescents; Obese adolescents; Obesity prevention program; Social media reminders; Effectiveness evaluation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Education group (Experimental): The group that will receive only an eight-week "Obesity Prevention Program."
  Interventions: Behavioral: Obesity prevention program
- Education + Social media supported group (Experimental): The group that will receive only an eight-week "Obesity Prevention Program." For 12 weeks after the program, supportive and reminder messages on the topic will be sent three days a week via social media networks.
  Interventions: Behavioral: Obesity prevention program; Behavioral: Social media messages
- Control group (No Intervention): No intervention will be made by the researcher during the study. Only data collection will be conducted. At the end of the study, the "Obesity Prevention Program" will be provided.

INTERVENTIONS:
Behavioral: Obesity prevention program — The Obesity Prevention Program was developed based on a literature review. Expert opinions (Public Health Nursing, Pediatric Nursing, Physical Therapy and Rehabilitation, Nutrition and Dietetics) were obtained for the educational content, and the final version was formulated. The training program is planned in eight sessions. The program will be scheduled at times convenient for students after prior discussion with the school administration. Two sessions per week will be conducted, with each session expected to last approximately 30-40 minutes. Students will utilize school computers and projectors during the training. The program will include verbal presentations, PowerPoint slides, brainstorming, exercises, games, written and visual materials, video screenings, and Q&A sessions. Adolescents will try on weighted T-shirts of different weights, fruit plates will be distributed during sessions, and bookmarks, magnets, and brochures will be provided at the end of the sessions.
  Arms: Education + Social media supported group; Education group
Behavioral: Social media messages — In addition to the program, a total of 36 short messages will be sent three times a week to the Education + Social Media Supported group.
  Arms: Education + Social media supported group

SUMMARY:
Childhood overweight and obesity are defined as crises that adversely affect health and well-being, pave the way for various health problems in the future, and are increasingly prevalent worldwide. Obesity is a significant public health issue as it predisposes children and adolescents to lifelong diseases and contributes to increased mortality and morbidity in adulthood. Eating behavior irregularities and excesses during childhood and adolescence lead to deteriorating health and rising obesity incidence. This condition causes significant issues in the respiratory, endocrine, cardiovascular, digestive, and orthopedic systems while also creating psychological effects, such as weight-related dissatisfaction and social exclusion.

The dramatic increase in childhood obesity worldwide indicates that children's health habits have shifted over time. Effective lifestyle modifications and behavioral interventions focusing on healthy nutrition, physical activity, and stress management are essential for preventing and reducing obesity. Since children and adolescents spend most of their time in schools or extracurricular activities, schools play a crucial role in instilling healthy behaviors. Healthy eating habits established during adolescence often translate into sustainable lifestyle choices in adulthood, underscoring the importance of addressing obesity at an early stage.

Social media-supported awareness programs developed to prevent obesity can be an effective solution, especially for overweight and obese adolescents. Combatting obesity during childhood and adolescence is vital for reducing lifelong obesity risks and promoting overall health. Identifying and controlling risk factors associated with obesity are critical steps in improving individuals' quality of life.

Aim This study aims to evaluate the effectiveness of an obesity prevention program designed for overweight and obese adolescents and supported by social media reminders.

Significance In recent years, obesity has become a widespread public health issue affecting all age groups, including adolescents. Sedentary lifestyles and evolving living standards are considered primary contributors to this trend. Adolescents' awareness of obesity as a health issue and their adoption of healthy lifestyle habits are key components in fighting obesity. Particularly in school environments, promoting healthy eating habits and enhancing knowledge can effectively reduce obesity incidence.

This study seeks to assess adolescents' obesity status, eating addictions, nutritional literacy, and obesity awareness, thereby fostering healthy behavioral changes. The findings of this research are expected to fill gaps in the existing literature and guide future strategies in combating obesity.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Being classified as overweight or obese according to BMI classification
* Currently enrolled in a high school in the district
* Having parental consent to participate in the study
* Having no physical or mental disabilities or chronic illnesses (e.g., diabetes, metabolic syndrome, heart disease, etc.)
* Having a social media account
* Using the internet and owning a smartphone

Exclusion Criteria:

* Incomplete completion of the study data collection forms
* Withdrawal from participation in the study
* Transferring to another school during the intervention period
* Discontinuing internet and phone usage during the intervention period
* Developing a chronic illness during the intervention period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The Healthy Eating Attitude Scale | 5-6 month
  The scale was developed to measure attitudes toward healthy eating. It consists of 21 items, a five-point Likert scale, and 4 factors. These factors are named Information on Nutrition (IN), Emotion for Nutrition (EN), Positive Nutrition (PN), and Malnutrition (M). The lowest score that can be obtained from the scale is 21, and the highest score is 105. As the score on the scale increases, the attitude levels towards healthy eating also increase.
The Eating Behavior Similar to Addiction Scale | 5-6 month
  The scale consists of 15 items and two subscales: appetite impulse and low diet control. The scale follows a five-point Likert format and is evaluated based on the total score. Higher scores on the scale indicate more pronounced addictive-like eating behaviors. A reduction in these behaviors is expected after the program.
The Obesity Awareness Level Scale | 5-6 month
  The scale consists of 21 items and follows a four-point Likert structure. It comprises three subdimensions: Obesity Awareness (OA), Nutrition (N), and Physical Activity (PA). As the total score and the scores obtained from the subdimensions increase, the awareness level also increases.
The Adolescent Nutrition Literacy Scale | 5-6 month
  The scale consists of 22 items and three subdimensions. Seven items form the Functional Nutrition Literacy subdimension, six items form the Interactive Nutrition Literacy subdimension, and nine items form the Critical Nutrition Literacy subdimension. The scale is based on a five-point Likert system, where responses are given as follows: "1 = strongly disagree; 2 = disagree; 3 = neither agree nor disagree; 4 = agree; 5 = strongly agree." The scale allows a minimum score of 22 and a maximum score of 110, and as the total score increases, nutrition literacy also improves.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz Universty, Kumluca, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No